CLINICAL TRIAL: NCT04237818
Title: The Evaluation of Chenopodium Formosanum and Fagopyrum Esculentum Extract on Anti-aging Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH108-REC1-147
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-01

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Chenopodium Formosanum and Fagopyrum Esculentum Extract drink (Experimental)
  Interventions: Dietary Supplement: Chenopodium Formosanum and Fagopyrum Esculentum Extract drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 2 bottle (30 mL) per day for 56 days
  Arms: Placebo drink
Dietary Supplement: Chenopodium Formosanum and Fagopyrum Esculentum Extract drink — consume 2 bottle (30 mL) per day for 56 days
  Arms: Chenopodium Formosanum and Fagopyrum Esculentum Extract drink

SUMMARY:
To assess Chenopodium Formosanum and Fagopyrum Esculentum Extract on skin anti-aging

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 20-65 years old
* Subjects must read and sign the informed consent form after the study has been fully explained.
* Subjects are willing to cooperate and comply with all of the regulation during the trial.
* Subject should inform to investigator immediately if adverse effect is happened.
* Subjects are willing to avoid UV overexposure during the trial (include indoor tanning treatment).

Exclusion Criteria:

* Subjects who have known cosmetic, drug or food allergies.
* Subjects who have severe desquamation, tattoo, sunburn, peeling skin or other skin condition might impact measurement.
* Subjects with any physical condition judged by the researcher not to be eligible for this study.
* Subjects with uncontrollable physical condition such as high blood pressure, thyroid disease, diabetes, etc.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Those who are currently participating in other clinical trials or who have just concluded a clinical trial two weeks ago.
* Women who have started contraceptive or change current hormone contraceptive methods within 3 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
The change of skin moisture | Change from Baseline skin moisture at 8 weeks
  Corneometer® CM825 is utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® dual MPA 580 is utilized to measure skin elasticity (parameter R2). Units: μm penetration depth into the probe opening, expressed as curves
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  3D Full-Face Skin Analyzer IRV is utilized to measure wrinkles. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® combo - 20 MHz High Freq. Ultrasound probe is utilized to scan and analyze skin collagen density. Units: Intensity score
The change of skin tone | Change from Baseline skin tone at 8 weeks
  3D Full-Face Skin Analyzer IRV was utilized to measure skin tone. Units: arbitrary units
The change of skin brightness | Change from Baseline skin brightness at 8 weeks
  3D Full-Face Skin Analyzer IRV is utilized to measure skin brightness. Units: arbitrary units
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Mexameter® MX 18 is utilized to measure skin melanin index. Units: arbitrary Mexameter® units (0-999)
The change of skin L*a*b* value | Change from Baseline skin L*a*b* value at 8 weeks
  Color Spectrophotometer SCM-104/108 is utilized to measure skin L*a*b* value. Units: arbitrary units

SECONDARY OUTCOMES:
The change of transepidermal water loss (TEWL) | Change from Baseline TEWL at 8 weeks
  Tewameter® TM 300 is utilized to measure transepidermal water loss. Units: g/hm²
The change of skin texture | Change from Baseline skin texture at 8 weeks
  3D Full-Face Skin Analyzer IRV is utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 8 weeks
  3D Full-Face Skin Analyzer IRV is utilized to measure skin pores. Units: arbitrary units
The change of skin spots | Change from Baseline skin spots at 8 weeks
  3D Full-Face Skin Analyzer IRV is utilized to measure skin spots. Units: arbitrary units
The change of skin erythema level | Change from Baseline skin erythema level at 8 weeks
  Mexameter® MX 18 is utilized to measure skin erythema level. Units: arbitrary Mexameter® units (0-999)
Self-assessment questionnaire | 8 weeks
  Questionnaire is utilized to assess skin condition of the subjects. Units: score

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Prof., Principal Investigator — China Medical University, China; Po-Yuan Wu, Dr., Study Director — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taiwan